CLINICAL TRIAL: NCT02436395
Title: Comparison the Influence of the Povidone-iodine or the Normal Saline Cleaning the Incision for the Incidence of the Surgical Site Infections for Gastric Cancer Patients With Gastrectomy- Randomized Controlled Trial
Brief Title: Povidone-iodine and the Normal Saline Cleaning the Incision for the SSIs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jian-Kun Hu, Prof. of Gastrointestinal Surgery Department, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCH-GC-03
Record Dates: First submitted 2014-12-07; First posted 2015-05-06 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Surgical Site Infections; Gastric Cancer; Dehiscence of Laparotomy Wound
Keywords: gastric cancer; gastrectomy; laparotomy; SSIs; povidone-iodine; normal saline
MeSH Terms: conditions — Surgical Wound Infection; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (povidone-iodine group) (Experimental): The surgical incision is washed by the mixed solution with 400ml 9% normal saline and 100ml 5% povidone-iodine solution.
  We declare that we have no conflicts of interest.
  Interventions: Procedure: Group A (povidone-iodine wash the surgical incision)
- Group B (normal saline group) (Experimental): The surgical incision is washed by the 500ml 0.9% normal saline.
  We declare that we have no conflicts of interest.
  Interventions: Procedure: Group B (normal saline wash the surgical incision)

INTERVENTIONS:
Procedure: Group A (povidone-iodine wash the surgical incision) — Gastric cancer patients underwent conventional open D2 total or subtotal gastrectomy and with povidone-iodine wash the surgical incision
  Arms: Group A (povidone-iodine group)
Procedure: Group B (normal saline wash the surgical incision) — Gastric cancer patients underwent conventional open D2 total or subtotal gastrectomy and with normal saline wash the surgical incision
  Arms: Group B (normal saline group)

SUMMARY:
Surgical site infections (SSIs) is one of the most common complications of upper abdominal surgery. Previous studies found that type of surgical incision, emergency operation or not, surgical duration, age of patient, body mass index, malignance duration, malnutrition, complications (diabetes, shock, anemia et al) and drug (Long-term use of corticosteroids) are closely associated with the incidence of SSIs. The general incidence rate of SSIs was about 5% to 40%, although using the preoperative skin disinfectant and other methods to prevent and reduce the SSIs. And for the gastrointestinal surgery, due to the potential risk of infection, SSIs is an important problem which cannot be ignored. On the other hand, gastric cancer is one of the most common digestive system tumors, and gastrectomy is the primary therapeutic options. Therefore, it is important to compare the whether the different liquid (1% povidone-iodine solution or the 0.9% normal saline) wash the incision can influent the incidence of the SSIs.

DETAILED DESCRIPTION:
Standard Operating Procedure (SOP)

1. Preoperative evaluation Patients satisfied with inclusion/exclusion criteria will be informed to join in the clinical study and signature the inform consent.
2. Randomization: Preoperative evaluation found that total or subtotal gastrectomy can be performed, the case will entrance into the Randomization period. Random numbers are computer-generated, with the third party applications.
3. Procedures: The surgical treatments is adopted the conventional open total or subtotal gastrectomy according to the Japanese Gastric Cancer treatments guidelines, 2010, Version 3. Patients in the Group A using the mixed solution with 400ml,0.9% normal saline and 100 ml，5%, povidone-iodine solution， and patients in the Group B with 500ml 0.9% normal saline solution to wash the abdominal surgical incision.
4. Postoperative recovery: Postoperative recovery period need to collect those relevant parameters of all the patients. All the relevant parameters had definitely definition in the Case Report Form of this study which included the preoperative, intraoperative and postoperative clinicopathologic characteristics.
5. Follow-up: Follow-up will last to the 30-day of the postoperative period. The postoperative complications is graded by the Clavien-Dindo classification. And the surgical site infections are the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed gastric adenocarcinoma, and predictively feasible of conventional open total gastrectomy or subtotal gastrectomy;
2. Predictively resectable diseases, of preoperative staging JGCA 14th Edition cT1N0M0-T4aN+M0, Ia-IIIc stage
3. Age：≤75 years, or ≥18 years;
4. Without serious disease and malignance disease;
5. WHO performance score ≤2, ASA score ≤3;
6. No limit to sexual and race;
7. Informed consent required.

Exclusion Criteria:

1. Emergence operation, because of obstruction, perforate, acute hemorrhage and et al;
2. Patients with laparoscopic or laparoscopic-assisted gastrectomy
3. Patients with other severe complications cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc;
4. Patients treated with neoadjuvant chemotherapy or radiation therapy which might affect the efficacy observation;
5. Severity mental diseases;
6. Primary lesion cannot be resected in the pattern of transabdominal gastrectomy, but for Whipple's procedure, or with a transthoracic approach surgery;
7. After signature the Clinical trial agreement, patients and their agent will quit the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Superficial incisional surgical site infections | 30-day of postoperative duration
  The ceriteria for defining a surgical site infection adopt the defination of the Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee.Am J Infect Control. 1999;27(2):97-132; quiz 133-4; discussion 96.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, M.D. Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China